CLINICAL TRIAL: NCT00276692
Title: Phase II Study of Irinotecan (CPT-11) in Children and Adolescents With High Risk Ewing's Sarcoma
Brief Title: Irinotecan in Treating Patients With Newly Diagnosed Ewing's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-ET-2003-04; CDR0000454550 (Registry Identifier: PDQ (Physician Data Query)); EU-20582
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Sarcoma
Keywords: metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well irinotecan works in treating patients with newly diagnosed Ewing's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the responsiveness of single-agent irinotecan hydrochloride in a patient population with newly diagnosed high-risk Ewing's sarcoma.

OUTLINE: This is an open-label, multicenter study.

Patients receive irinotecan hydrochloride IV over 1 hour on day 1. Treatment repeats every 21 days for 2 courses. After completion of 2 courses of therapy, patients may receive additional treatment at the discretion of the treating physician.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Ewing's tumor

  * Ewing's sarcoma or peripheral primitive neuroectodermal tumor of bone or soft tissue
  * High-risk disease (R3), defined as metastases at extrapulmonary/pleural sites
* Newly diagnosed disease
* Measurable primary and/or metastatic disease

  * At least one bidimensionally measurable lesion
* Concurrent enrollment on EURO-Ewing99 clinical trial required

PATIENT CHARACTERISTICS:

* No abnormal cardiac function, including any of the following:

  * Fractional shortening < 29%
  * Ejection fraction < 40%
* Glomerular filtration rate ≥ 60mL/min
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No prior or current history of chronic diarrhea, bowel obstruction, sub obstruction, Crohn's disease, or ulcerative colitis
* No other medical, psychiatric, or social condition incompatible with the study treatment

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No more than 45 days since prior definitive biopsy

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Response as measured by MRI following course 2

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Morland, MD, Study Chair — Birmingham Children's Hospital
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales